CLINICAL TRIAL: NCT02491879
Title: Ketoprofen Gel vs Placebo in Patients Presented With Low-back Pain to Emergency Department: A Ranodmized Controlled Trial
Brief Title: Ketoprofen Gel vs Placebo in Low Back Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Collaborators: Kocatepe University (Other); Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24924
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Mechanical Low Back Pain
Keywords: mechanical low back pain; emergency department; ketoprofen; gel
MeSH Terms: conditions — Low Back Pain; Emergencies | interventions — Ketoprofen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen (Experimental): Ketoprofen gel
  Interventions: Drug: Ketoprofen
- Placebo (Placebo Comparator): Placebo form of ketoprofen gel
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketoprofen — 2.5% Ketoprofen gel with a 2 g local use
  Other Names: Fastjel
  Arms: Ketoprofen
Other: Placebo — Placebo gel with a 2 g local use
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
This study aimed to analyse the analgesic effect of ketoprofen gel in patients presented with mechanical low-back pain to the emergency department.

DETAILED DESCRIPTION:
Mechanical low-back pain which warrants immediate pain relief is not an infrequent symptom for emergency department physicians to deal with. Parenteral analgesic is the most common drugs for the these patients in emergency department. However, pain killers in gel forms have not been studied sufficiently for ceasing the pain of these patients. This study aimed to analyse the analgesic effect of ketoprofen gel in patients presented with mechanical low-back pain to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and lower 65 years old
* Patients presented with mechanical low-back pain

Exclusion Criteria:

* Pain more than 24 hours
* Pain lower than with a pain score of 40 mm
* Allergy to ketoprofen
* Drug or alcohol addiction
* pregnancy and breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 30 minutes
  Pain reduce will be measured by visual analogue scale score at 30 minutes

SECONDARY OUTCOMES:
Adverse outcome | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, MD, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)